CLINICAL TRIAL: NCT02253199
Title: The Effect of Age on the Median Effective Dose (ED50) of Intranasal Dexmedetomidine for Rescue Sedation Following Failed Sedation With Oral Chloral Hydrate During Magnetic Resonance Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Wenhua Zhang, Director, Clinical Resesearch, Guangzhou Women and Children's Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double
Other Study IDs: WZhang-02
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Aged; Drug; Dose-Response Relationship

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1-6 months (Group 1) (Active Comparator): Subjects stratified into four groups according to age: 1-6 months (Group 1), 7-12 months (Group 2),13-24 months (Group 3), 26-36 months (Group 4).
  Interventions: Drug: intranasal dexmedetomidine
- 7-12 months (Group 2) (Active Comparator): Subjects stratified into four groups according to age: 1-6 months (Group 1), 7-12 months (Group 2),13-24 months (Group 3), 26-36 months (Group 4).
  Interventions: Drug: intranasal dexmedetomidine
- 13-24 months (Group 3) (Active Comparator): Subjects stratified into four groups according to age: 1-6 months (Group 1), 7-12 months (Group 2),13-24 months (Group 3), 26-36 months (Group 4).
  Interventions: Drug: intranasal dexmedetomidine
- 25-36 months (Group 4) (Active Comparator): Subjects stratified into four groups according to age: 1-6 months (Group 1), 7-12 months (Group 2),13-24 months (Group 3), 26-36 months (Group 4).
  Interventions: Drug: intranasal dexmedetomidine

INTERVENTIONS:
Drug: intranasal dexmedetomidine — Children who were not adequately sedated ( no evidence of adequate sedation within 30 min after administration of Initial dose of chloral hydrate) received a bolus of intranasal dexmedetomidine which adjusted by the "Dixon up-and-down method for rescue sedation.
  The first child received 0.8mcg/Kg of intranasal dexmedetomidine dose (100mcg/ml), and the dose interval was set at 0.1mcg/Kg.

SUMMARY:
Increasing evidences suggest that dexmedetomidine Pharmacokinetic are different in children. We performed a up-down sequential allocation study to determine the ED50 for rescue sedation following sedation failures in children and to investigate age-related differences in the rescue sedation with dexmedetomidine.

DETAILED DESCRIPTION:
About 150 children who were not adequately sedated ( no evidence of adequate sedation within 30 min after administration of Initial dose of chloral hydrate) were stratified into four age groups as follows: 1-6 month, 7 -12 month, 13 -24 month, and 25-36 month. The intranasal dexmedetomidine dose was determined by the success or failure of rescue sedation achieved by the previous patients, according to Dixon's up-down sequential allocation method. Successful sedation was defined as a MOAA/S(modified Observer Assessment of Alertness and Sedation) of between 0 and 3. The EC50 were estimated from the up-and-down sequences using the method of Dixon and Massey and logistic regression. Patients' sedation status, sedation induction time, time to Wake up, blood pressure, heart rate, and oxygen saturation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* 150 children of ASA physical status I or II, aged between 1 and 36 months, failed chloral hydrate sedation during MRI scanning,

Exclusion Criteria:

* known allergy or hypersensitive reaction to drugs of this study, Weight greater than 20 kg or less than 4.5 kg, organ dysfunction, pneumonia, acute upper respiratory airway inflammation, preterm, cardiac arrhythmia and congenital heart disease.

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The median effect dose of intranasal dexmedetomidine | up to 1 hours after MRI scaning
  Sedation status was evaluated by a attending anesthesiologists every 5-10 min with a 6-point sedation scale, which was modified from the Modified Observer Assessment of Alertness and Sedation Scale (MOAA/S).successful sedation was defined as an MOAA/S of between 0 and 3

SECONDARY OUTCOMES:
sedation induction time | up to 30 min after rescue drug administration
  Successful sedation was defined as an MOAA/S of between 0 and 3, and sedation induction time was defined as the time from rescue drug administration to the onset of satisfactory sedation
  0 Does not respond to a noxious stimulus
  1. Does not respond to mild prodding or shaking
  2. Responds only after mild prodding or shaking
  3. Responds only after name is called loudly orrepeatedly
  4. Lethargic response to name spoken in normal tone
  5. Appears asleep, but responds readily to namespoken in normal tone
  6. Appears alert and awake, responds readily to namespoken in normal tone
Wake -up time | up to 4 hours after rescue drug administration
  Children were classified as awake if the MOAA/S was between 4 and 6. Wake -up time was defined as the time from successful sedation until the time that the child awoke

OTHER OUTCOMES:
heart rate | baseline, before and 15 , 60, 75, 90 min after rescue drug administration
  changes in heart rates at the baseline, before and 15 , 60, 75, 90 min after rescue drug administration
non-invasive systolic blood pressure | baseline, before and 15 , 60, 75, 90 min after rescue drug administration
  changes in the non-invasive systolic blood pressure at the baseline, before and 15 , 30, 60, 75, 90 min after rescue drug administration
Oxyhemoglobin desaturation | baseline and four hours after rescue medicine administration
  Significant Oxyhemoglobin desaturation was defined as<94%

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology of Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang W, Fan Y, Zhao T, Chen J, Zhang G, Song X. Median Effective Dose of Intranasal Dexmedetomidine for Rescue Sedation in Pediatric Patients Undergoing Magnetic Resonance Imaging. Anesthesiology. 2016 Dec;125(6):1130-1135. doi: 10.1097/ALN.0000000000001353. PMID 27627818